CLINICAL TRIAL: NCT00745186
Title: A Randomized, Open Label, Four Way Crossover Study to Compare the Pharmacokinetics, Pharmacodynamics and Safety After Intramuscular (IM) Administration of Mayne Glucagon for Injection With Glucagen® (Novo Nordisk) in Healthy Volunteers.
Brief Title: Pharmacokinetics (PK) and Pharmacodynamics (PD) of Mayne Glucagon for Injection Compared With Glucagen® (Novo Nordisk) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GLC061
Record Dates: First submitted 2008-09-02; First posted 2008-09-03 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2015-06

CONDITIONS: Hypoglycemia
MeSH Terms: conditions — Hypoglycemia | interventions — Glucagon-Like Peptide 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Glucagen
  Interventions: Drug: Glucagen
- 2 (Experimental): Mayne Glucagon
  Interventions: Drug: Mayne Glucagon

INTERVENTIONS:
Drug: Glucagen — 0.2 mg or 1 mg Glucagen single injection
  Arms: 1
Drug: Mayne Glucagon — 0.2 mg or 1 mg Mayne Glucagon
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics and pharmacodynamic bioequivalence and safety of Hospira Glucagon for Injection and GlucaGen® in healthy volunteers.

DETAILED DESCRIPTION:
Glucagon has been shown to be effective in the treatment of hypoglycemia, low blood sugar levels, in patients with diabetes. It primarily functions as a counter-regulatory hormone by opposing the actions of insulin to maintain blood glucose levels. A major problem for diabetic patients with hypoglycemia is the development of defective counter regulatory responses including reduced or absent glucagon responses to hypoglycemia. Mayne Glucagon for Injection has been developed as an alternative to currently marketed products.

Administration of exogenous glucagon i.e., not produced in the body, has been shown to be effective in the treatment of low blood sugar in patients with diabetes. Mayne has developed a product, Glucagon for Injection, which is an alternative to currently marketed products. The only difference is the source of the active ingredient. The formulation, routes of administration, dosage regimen and indications of Mayne Glucagon for Injection are identical to those currently registered for the marketed product.

A total of 28 healthy volunteers will be recruited into this study at one investigational site.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Male or female aged 18-50 years inclusive
* Body weight between 50 - 100 kg and body mass index (BMI) between 18 and 30 kg/m2 or, if outside the range, considered not clinically significant by the investigator
* Non-smokers or ex-smokers who have not smoked with in the previous 3 months
* Written informed consent given
* Willing and able to comply with the requirements of the protocol and available for the planned duration of the study
* Subject must agree to use an adequate method of contraception during the study and for 12 weeks after the last dose of investigational medicinal product (IMP). Adequate methods of contraception for subject or partner include condoms with spermicide gel, diaphragm with spermicide gel, coil (intrauterine device), surgical sterilisation, subdermal implant, vasectomy, oral contraceptive pill, depot progesterone injections and abstinence. If a volunteer is usually not sexually active but becomes active he/she or their partner must use one of the contraceptive methods listed . Male subjects whose partner is of child bearing potential must ensure that they or their partner use effective contraception for the course of the study and 12 weeks thereafter

Exclusion Criteria:

* History or presence of any clinically significant findings that, in the opinion of the investigator, would preclude inclusion in the study
* History or presence of clinical significant gastrointestinal pathology or symptoms, liver or kidney disease or any other condition that might interfere with the absorption, distribution, metabolism or excretion of the drug.
* Any clinically significant laboratory findings
* Clinically significant abnormalities in 12-lead electrocardiogram (ECG) results
* Positive pregnancy test or lactation
* Participation in any other clinical study using an investigational product or device within the previous 12 weeks
* Positive human immunodeficiency virus (HIV), Hepatitis B or C test
* History of drug or alcohol abuse within the past two years or alcohol consumption greater than 21 units per week for males and greater than 14 units per week for females
* Blood donation of ≥ 500 mL in the previous 12 weeks
* Hypersensitivity to Glucagon and/or any excipients
* Use of prescription medicines or St John's Wort in the previous 2 weeks. The use of over-the-counter medicines within 5 days of dosing except those deemed by the investigator not to interfere with the outcome of the study. Vitamins, minerals and nutritional supplements may be taken at the discretion of the investigator. Hormonal contraceptives will be permitted.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2007-08; Primary Completion 2007-10 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve from Time 0 to the Last Time Point (AUC0-tlast) for 1 mg Dose Level | Pre-dose: 20, 10 and 5 min; Post-dose: 5, 10, 15, 20, 25, 30, 35, 40, 45, 60, 90, 120, 150, 180 and 240 minutes.
Maximum Glucagon Concentration Observed (Cmax) for 1 mg Dose Level | Pre-dose: 20, 10 and 5 min; Post-dose: 5, 10, 15, 20, 25, 30, 35, 40, 45, 60, 90, 120, 150, 180 and 240 minutes.
Maximum Blood Glucose Concentration Observed (BG Cmax) for 1 mg Dose Level | Pre-dose: 20, 10 and 5 min; Post-dose: 5, 10, 15, 20,25,30, 35, 40, 45, 60, 90, 120, 150, 180 and 240 minutes.

SECONDARY OUTCOMES:
Area under the curve from time 0 extrapolated to infinity (AUC0-inf) for 1 mg Dose Level | Pre-dose: 20, 10 and 5 min; Post-dose: 5, 10, 15, 20, 25, 30, 35, 40, 45, 60, 90, 120, 150, 180 and 240 minutes.
Time at which Cmax occurs (Tmax) for 1 mg Dose Level | Pre-dose: 20, 10 and 5 min; Post-dose: 5, 10, 15, 20, 25, 30, 35, 40, 45, 60, 90, 120, 150, 180 and 240 minutes.
Elimination half life (T1/2) for 1 mg Dose Level | Pre-dose: 20, 10 and 5 min; Post-dose: 5, 10, 15, 20,25, 30, 35, 40, 45, 60, 90, 120, 150, 180 and 240 minutes.
Area Under the Curve from Time 0 to the Last Time Point (AUC0-tlast) for 0.2 mg Dose Level | Pre-dose: 20, 10 and 5 min; Post-dose: 5, 10, 15, 20, 25, 30, 35, 40, 45, 60, 90 and 120 minutes.
Maximum Glucagon Concentration Observed (Cmax) for 0.2 mg Dose Level | Pre-dose: 20, 10 and 5 min; Post-dose: 5, 10, 15, 20, 25, 30, 35, 40, 45, 60, 90 and 120 minutes.
Area under the curve from time 0 extrapolated to infinity (AUC0-inf) for 0.2 mg Dose Level | Pre-dose: 20, 10 and 5 min; Post-dose: 5, 10, 15, 20, 25, 30, 35, 40, 45, 60, 90 and 120 minutes.
Time at which Cmax occurs (Tmax) for 0.2 mg Dose Level | Pre-dose: 20, 10 and 5 min; Post-dose: 5, 10, 15, 20, 25, 30, 35, 40, 45, 60, 90 and 120 minutes.
Elimination half-life (T1/2) for 0.2 mg Dose Level | Pre-dose: 20, 10 and 5 min; Post-dose: 5, 10, 15, 20, 25, 30, 35, 40, 45, 60, 90 and 120 minutes.
Time at which Blood Glucose Cmax occurs (BG Tmax) for 1 mg Dose Level | Pre-dose: 20, 10 and 5 min; Post-dose: 5, 10, 15, 20, 25, 30, 35, 40, 45, 60, 90, 120, 150, 180 and 240 minutes.
Area under the curve from time 0 to return to baseline (rtb) for 1 mg Dose Level | Pre-dose: 20, 10 and 5 min; Post-dose: 5, 10, 15, 20, 25, 30, 35, 40, 45, 60, 90, 120, 150, 180 and 240 minutes.
Maximum absolute Blood Glucose excursion (MAE) from baseline for 1 mg Dose Level | Pre-dose: 20, 10 and 5 min; Post-dose: 5, 10, 15, 20, 25, 30, 35, 40, 45, 60, 90, 120, 150, 180 and 240 minutes.
Area under the glucose excursion versus time curve from 0 to rtb for 1 mg Dose Level | Pre-dose: 20, 10 and 5 min; Post-dose: 5, 10, 15, 20, 25, 30, 35, 40, 45, 60, 90, 120, 150, 180 and 240 minutes.
The earliest recorded time of the MAE for 1 mg Dose Level | Pre-dose: 20, 10 and 5 min; Post-dose: 5, 10, 15, 20, 25, 30, 35, 40, 45, 60, 90, 120, 150, 180 and 240 minutes.
Maximum Blood Glucose Concentration Observed (BG Cmax) for 0.2 mg Dose Level | Pre-dose: 20, 10 and 5 min; Post-dose: 5, 10, 15, 20, 25, 30, 35, 40, 45, 60, 90 and 120 minutes.
Time at which Blood Glucose Cmax occurs (BG Tmax) for 0.2 mg Dose Level | Pre-dose: 20, 10 and 5 min; Post-dose: 5, 10, 15, 20, 25, 30, 35, 40, 45, 60, 90 and 120 minutes.
Area under the curve from time 0 to return to baseline (rtb) for 0.2 mg Dose Level | Pre-dose: 20, 10 and 5 min; Post-dose: 5, 10, 15, 20, 25, 30, 35, 40, 45, 60, 90 and 120 minutes.
Maximum absolute Blood Glucose excursion (MAE) from baseline for 0.2 mg Dose Level | Pre-dose: 20, 10 and 5 min; Post-dose: 5, 10, 15, 20, 25, 30, 35, 40, 45, 60, 90 and 120 minutes.
Area under the glucose excursion versus time curve from 0 to rtb for 0.2 mg Dose Level | Pre-dose: 20, 10 and 5 min; Post-dose: 5, 10, 15, 20, 25, 30, 35, 40, 45, 60, 90 and 120 minutes.
The earliest recorded time of the MAE for 0.2 mg Dose Level | Pre-dose: 20, 10 and 5 min; Post-dose: 5, 10, 15, 20, 25, 30, 35, 40, 45, 60, 90 and 120 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Mair, Principal Investigator — Syneos Health
Locations (1):
- Charles River Laboratories, Edinburgh, United Kingdom